CLINICAL TRIAL: NCT07101731
Title: The Effects of Hypopressive Exercises on Urinary Incontinence and Erectile Dysfunction After Radical Prostatectomy: A Randomized Controlled Trial
Brief Title: Effects of Hypopressive Exercises on Urinary Incontinence and Erectile Dysfunction After Radical Prostatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Betül ERBAY, Lecturer, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBU-RPHEE-2025-01
Record Dates: First submitted 2025-07-18; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer (Post Prostatectomy); Urinary Incontinence; Erectile Dysfunction Following Radical Prostatectomy; Pelvic Floor Muscle Training
Keywords: Radical Prostatectomy; Urinary Incontinence; Erectile Dysfunction; Pelvic Floor Muscle Training; Hypopressive Exercises
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence; Erectile Dysfunction

STUDY DESIGN:
Masking Description: No masking was performed due to the nature of the intervention. Participants and investigators were aware of the group assignments. türkçesi
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Floor Home Exercise + Supervised Hypopressive Exercise Group (Experimental): Participants will perform daily home-based pelvic floor muscle exercises and also attend supervised hypopressive exercise sessions twice a week for 8 weeks.
  Interventions: Behavioral: Pelvic Floor Muscle Training (PFMT); Behavioral: Hypopressive Exercises
- Pelvic Floor Home Exercise Only Group (Active Comparator): Participants will be instructed to perform home-based pelvic floor muscle exercises daily for 8 weeks. No supervised exercise sessions will be provided.
  Interventions: Behavioral: Pelvic Floor Muscle Training (PFMT)

INTERVENTIONS:
Behavioral: Pelvic Floor Muscle Training (PFMT) — Participants in the control group will receive an individualized home-based pelvic floor muscle exercise program. Exercises will be performed once daily for 8 weeks, focusing on voluntary pelvic floor contractions in various positions (supine, sitting, standing). Participants will receive initial training and written instructions from a physiotherapist, and will be contacted weekly to monitor adherence.
Behavioral: Hypopressive Exercises — Participants in the experimental group will attend supervised hypopressive exercise sessions twice per week for 8 weeks. These sessions involve specific postural sequences combined with breathing and apnea techniques aimed at reducing intra-abdominal pressure while activating pelvic floor and abdominal muscles. Sessions will be led by a physiotherapist and adapted based on individual performance and posture tolerance.
  Arms: Pelvic Floor Home Exercise + Supervised Hypopressive Exercise Group

SUMMARY:
This randomized controlled trial investigates the effects of hypopressive exercises on urinary incontinence and erectile dysfunction in men following radical prostatectomy. Participants will be randomly assigned to one of two groups: a control group receiving home-based pelvic floor muscle exercises and an experimental group receiving both pelvic floor muscle exercises and supervised hypopressive exercises twice per week. The study aims to determine whether the addition of hypopressive techniques, which target coordinated activation of the pelvic floor and abdominal muscles without increasing intra-abdominal pressure, offers greater improvements in urinary and sexual function. Primary outcomes include pelvic floor muscle strength and endurance, while secondary outcomes include urinary incontinence severity, erectile function, and quality of life.

DETAILED DESCRIPTION:
Prostate cancer is one of the most common malignancies among men, with radical prostatectomy being a widely used treatment option. However, post-surgical complications such as urinary incontinence and erectile dysfunction significantly affect the quality of life of these patients. Pelvic floor muscle training (PFMT) is frequently recommended to manage these complications, yet its standalone effectiveness remains debatable.

Recent literature highlights that optimal pelvic floor function is achieved through coordinated activation with abdominal and respiratory muscles, such as the transversus abdominis, rectus abdominis, and diaphragm. Despite this, conventional PFMT protocols for post-prostatectomy patients often neglect this integrated muscle synergy. Hypopressive exercises, which involve postural techniques with apnea and breathing control, have been shown to activate both pelvic floor and abdominal muscles without increasing intra-abdominal pressure.

This study aims to evaluate the effects of hypopressive exercises, in addition to standard pelvic floor exercises, on pelvic floor muscle strength, urinary incontinence severity, and erectile function in post-prostatectomy men. The study will be conducted with two arms: a control group performing home-based pelvic floor exercises and an experimental group performing the same PFMT along with supervised hypopressive exercises twice weekly for 8 weeks. Outcomes will be assessed pre- and post-intervention, focusing on both physical performance and patient-reported measures.

ELIGIBILITY:
Inclusion Criteria

* Male individuals diagnosed with prostate cancer who have undergone radical prostatectomy
* Experiencing both urinary incontinence and erectile dysfunction
* Age > 55 years
* A score of 24 or higher on the Mini-Mental State Examination (MMSE)
* Literate (able to read and write)
* Willingness to participate in the study (signed informed consent)
* Ability to voluntarily contract pelvic floor muscles
* Ability to cooperate with the assessments and interventions used in the study

Exclusion Criteria

* History of urinary incontinence before surgery
* Congenital abnormalities of the urinary system
* Presence of neurological disorders
* History of transurethral resection of the prostate (TURP)
* Diagnosis of chronic obstructive pulmonary disease (COPD) and/or chronic restrictive pulmonary disease
* History of inguinal hernia
* Previous or current history of radiation therapy
* Surgical or postoperative complications that prevent early physiotherapy intervention (e.g., urinary tract infection, bladder neck stenosis)

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in urinary incontinence severity measured by 1-hour Pad Test | Baseline and 8 weeks
  The 1-hour Pad Test, standardized by the International Continence Society (ICS), will be used to objectively assess urinary leakage. A weight gain of >1g indicates a positive test. Severity will be classified as mild (<2g), moderate (2-10g), severe (10-50g), or very severe (>50g). The difference in pad weight pre- and post-intervention will be recorded.
Change in pelvic floor muscle strength measured by Modified Oxford Scale | Baseline and 8 weeks
  Pelvic floor muscle strength will be assessed by manual digital palpation in a side-lying position with knees flexed at 45 degrees. Strength will be scored using the Modified Oxford Scale, which ranges from 0 (no contraction) to 5 (strong contraction). Higher scores indicate better pelvic floor muscle strength.
Change in pelvic floor muscle endurance measured in seconds | Baseline and Week 8
  Pelvic floor muscle endurance will be assessed by instructing participants to sustain a maximal voluntary pelvic floor muscle contraction for as long as possible in a side-lying position with knees flexed at 45 degrees. The duration (in seconds) for which the contraction is maintained without loss of force will be recorded. Longer durations indicate greater endurance.

SECONDARY OUTCOMES:
Change in erectile function measured by IIEF-5 | Baseline and 8 weeks
  Erectile function will be assessed using the 5-item version of the International Index of Erectile Function (IIEF-5). Total scores range from 5 to 25, with lower scores indicating more severe erectile dysfunction. The change in total score from baseline to post-intervention will be analyzed.
Change in urinary incontinence severity and impact measured by ICIQ-SF | Baseline and 8 weeks
  The International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) will be used to assess perceived severity and quality of life impact of urinary incontinence. The total score is based on responses to questions 3, 4, and 5 (range: 0-21). Higher scores indicate more severe incontinence.
Change in quality of life measured by King's Health Questionnaire | Baseline and 8 weeks
  The King's Health Questionnaire will be used to assess health-related quality of life in individuals with urinary incontinence. The questionnaire includes multiple subdomains, with scores ranging from 0 (best health status) to 100 (worst). A decrease in score indicates improvement.
Change in urinary frequency and incontinence episodes measured by 3-day bladder diary | Baseline and 8 weeks
  A 3-day bladder diary will be used to document frequency of urination, incontinence episodes, and fluid intake. Data from weekdays and weekends will be averaged to calculate daily means. Change in urination and leakage frequency from baseline to Week 8 will be analyzed.
Change in perceived urinary symptom severity measured by Patient Global Impression of Severity (PGI-S) | Baseline and 8 weeks
  Participants will rate the perceived severity of urinary incontinence using the Patient Global Impression of Severity (PGI-S) scale. The PGI-S is a 4-point scale ranging from 1 (normal) to 4 (severe). Higher scores indicate worse perceived urinary symptom severity. Change in score from baseline to Week 8 will be used to evaluate subjective symptom burden.
Perceived improvement in urinary symptoms measured by Patient Global Impression of Improvement (PGI-I) | Week 8
  Participants will evaluate the overall change in their urinary symptoms using the Patient Global Impression of Improvement (PGI-I) scale. The PGI-I is a 7-point scale ranging from 1 (very much better) to 7 (very much worse). Lower scores indicate greater perceived improvement. This measure will be used to assess subjective global change in urinary symptoms after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Gülhane Training and Research Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data (IPD) sharing decision has not been finalized. Although publication of the study results is planned, the possibility of sharing de-identified IPD with other researchers will depend on institutional policies, ethical approvals, and publication guidelines.